CLINICAL TRIAL: NCT05552599
Title: The Effect of Body Temperature Changes Durıng Total Knee Arthroplasty Surgery on The Formatıon of Early Postoperatıve Pressure Sore
Brief Title: Body Temperature Changes and Early Postoperatıve Pressure Sore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Zehra UNAL, Principal Investigator, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HititZ
Record Dates: First submitted 2022-07-04; First posted 2022-09-23 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Pressure Sore; Orthopedic Disorder; Hypothermia; Nursing Caries
MeSH Terms: conditions — Pressure Ulcer; Musculoskeletal Diseases; Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- woolen blanket (Experimental): Preoperative pressure sore risk was assessed with the Braden Risk Assessment Scale. The patient's room temperature was recorded on the day of surgery before the patient was admitted for the operation. Body temperature was measured before the patient wore surgical gown. Before leaving the room, patient's body was covered with a woolen blanket. The temperature of the operating room was recorded. Body temperature was stabilized under normothermic conditions with a woolen blanket until the operation began. Body temperature was measured before anesthesia was given. Body temperature was measured in the 1st, 2nd and 3rd hour after anesthesia was given. The patient was evaluated with the Braden Risk Assessment Scale on the first, second and third postoperative days.
  Interventions: Procedure: woolen blanket
- standard of care (No Intervention): Preoperative pressure sore risk was assessed with the Braden Risk Assessment Scale. The patient's room temperature was recorded on the day of surgery before the patient was taken to the operation. Body temperature was measured before the patient wore surgical clothes. The temperature of the operating room was recorded. Body temperature was measured before anesthesia was givenBody temperature was measured at the 1st, 2nd and 3rd hour after anesthesia was given. The patient was evaluated with the Braden Risk Assessment Scale on the first, second and third postoperative days.

INTERVENTIONS:
Procedure: woolen blanket — Woolen blanket: The people in the experimental group were treated with a standard hospital woolen.
  Arms: woolen blanket

SUMMARY:
This study aims to determine effect of body temperature changes during total knee arthroplasty surgery on early postoperative pressure sore formation.

DETAILED DESCRIPTION:
BACKGROUND: Intraoperative hypothermia for a prolonged period increases the risk of hospital-acquired pressure sores.

PURPOSE: This study aims to determine effect of body temperature changes during total knee arthroplasty surgery on early postoperative pressure sore formation.

METHODS: This experimental study was performed with experimental-control group (N=122) patients. Data were collected with "Personal Information Form", "Body and Ambient Temperature Record Form", "Braden Risk Assessment Scale". Experimental group participants were covered with a wool blanket, and control group was given standard care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-85 years
* Hospitalized for at least four days and accepted to participate were included in the study.

Exclusion Criteria:

* Under the age of 20 - over 85,
* Pregnant and having comorbid diseases,
* Spinal cord injuries,
* Skin problems in areas where there is a risk of pressure loss,
* Undergoing hemodialysis,
* Having creatinine and serum albumin levels higher than 3 mg/dl,
* Having immobility, incontinence, anemic, having malignant tumor(s),
* BMI <19 or BMI >40,
* Hemoglobin level below 10 g/dl,
* Infection,
* American Society of Anesthesiology (ASA) score of 3 or more,
* Experiencing friction, tearing and shearing,
* Undergoing more than one surgical intervention,
* Having conditions requiring the use of non-normal anesthetic agents and sedation,
* Using vasoconstrictive drugs,
* Using positioning devices,
* Undergoing prolonged surgical intervention,
* Having arterial pressure lower than 32 mmHg,
* Having diabetes mellitus requiring insulin therapy.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2019-03-03 (Actual); Study Completion 2019-03-03 (Actual)

PRIMARY OUTCOMES:
In collecting the data, three different data collection tools were used: "Personal Information Form" | 12 months
  The personal information form prepared by the researcher using the literature consisted of seven items in total, questioning age, gender, marital status, educational status, occupational status, income level and previous hospitalization experience.
Body and Ambient Temperature Record Form" | 12 months
  It is the form that allows to keep track of the temperature of the patient's room, the temperature of the patient's body before putting on the surgical gown, the temperature of the operating room, the body temperature before anesthesia, and the body temperature in the first, second and third hours following anesthesia.
"Braden Risk Assessment Scale". | 12 months
  Braden Risk Assessment Scale includes six sub-scales: sensory perception, moisture, activity, mobility, nutrition, friction and shear.
  The total score of the scale ranges between 6-23. A total score of 12 or lower shows high risk; 13-14 moderate risk; 15-16 low risk, and 15-18 considered mild risk for people over 75 years old. The scale includes six sub-scales: sensory perception, moisture, activity, mobility, nutrition, friction and shear. The sub-scales of sensory perception, moisture, activity, mobility and nutrition are scored 1-4; the friction-shear sub-scale 1-3, and the total score ranges between 6-23. The risk increases as the total score decreases. 15-18 points are accepted as low risk in people over 75 years old.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra UNAL, Principal Investigator — zehra86_sevgi@hotmail.com
Locations (2):
- Turkey (Türkiye) (2):
  - Hitit University, Çorum
  - HititU, Çorum

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR